CLINICAL TRIAL: NCT05558189
Title: Vibrotactile Coordinated Reset for the Treatment of Post Surgery Refractory Parkinson's Disease Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Peter Tass, MD, PhD, Protocol Director, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 67601
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Vibrotactile Coordinated Reset (vCR) (Experimental): Vibrotactile Coordinated Reset delivers vibratory stimulation to the fingertips of each hand. A specific pattern of vibration to each fingertip is delivered which theoretically disrupts abnormal synchrony in the brain.
  Interventions: Device: Vibrotactile Coordinated Reset (vCR)

INTERVENTIONS:
Device: Vibrotactile Coordinated Reset (vCR) — The purpose of this study is to test the efficacy of vibrotactile coordinated reset stimulation on human subject participants who have refractory Parkinson's disease post surgical treatment

SUMMARY:
The purpose of our study is to evaluate Vibrotactile Coordinated Reset stimulation (vCR) and its effects on refractory post-surgery PD. vCR will be administered with a device called the Stanford Glove. vCR is expected to provide patients with a non-invasive alternative to the most widely used treatments such as levodopa and or deep brain stimulation. Patients will be followed for two years.

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of enrollment: 35 - 92 years
2. Diagnosis of idiopathic Parkinson's disease
3. Surgical treatment for Parkinson's disease that does not involve Deep Brain Stimulation
4. Fluent in English
5. Appropriate social support if required during an off state.
6. Comfortable with technology; can use a computer, check email, and access the internet; can initiate and engage in a virtual meeting for training and monitoring purposes.
7. Lives in the United States

Exclusion Criteria:

1. Any significant neuro-psychiatric problems, including acute confusional state, ongoing psychosis, or suicidal tendencies
2. Any current drug or alcohol abuse.
3. Participation in another drug, device, or biologics trial concurrently or within the preceding 30 days. Any other trial participation should be approved by the Principal Investigators.
4. Pregnancy, breast-feeding or wanting to become pregnant
5. Patient is unable to communicate properly with staff (i.e., severe speech problems)
6. Excessive drooling
7. Sensory abnormalities of the fingertips
8. Deep Brain Stimulation treatment
9. PD symptoms so severe and that the patient is bed-bound

Ages: 35 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-11-21 (Estimated); Study Completion 2026-11-21 (Estimated)

PRIMARY OUTCOMES:
Movement Disorders Society Unified Parkinson's Disease Rating Scale Part 3 (MDS-UPDRS III) change from baseline to 24 months. | 24 months
  This scale measures motor ability within Parkinson's patients. For part 3, the scales minimum values is 0 and max value is 132. Higher scores indicate more impaired motor ability, while lower scores indicate less impaired motor ability. A score of 0 indicates no motor impairment.

SECONDARY OUTCOMES:
Levodopa equivalent daily dose (LEDD) change from baseline to 24 months | 24 months
  LEDD is calculated as a daily sum of levodopa in each Parkinson's medication
Communicative Participation Item Bank (CPIB; Short Form) change from baseline to 24 months. | 24 months
  The CPIB is a questionnaire that measures speech complications. The questionnaire is scored from 0 to 30, with a higher score indicating increased speech difficulties.
Voice Handicap Index (VHI-10) change from baseline to 24 months | 24 months
  This questionnaire can be filled out by patients and assesses the impact that voice problems and limitations have on the individual's overall daily function. Questionnaire is scored from 0 to 40, with a higher score indicating increased speech difficulties.
Freezing of gait questionnaire (FOG) change from baseline to 24 months | 24 months
  The Freezing of Gait Questionnaire (FOG) assesses severity unrelated to falls in patients with Parkinson's Disease (PD), FOG frequency, disturbances in gait, and relationship to clinical features conceptually associated with gait and motor aspects (e.g., turning). The FOG is comprised of 6 questions measured on a 0 to 4 scale (where 0 is normal and 4 represents severe abnormalities). The scores are summed together with 0 representing the best possible score and 24 representing the worst possible score.
Vibratory temporal discrimination task (VTDT) change from baseline to 24 months. | 24 months
  The vibratory temporal discrimination task (VTDT) consists of two vibratory bursts, with one burst delivered to the index finger and one burst to the middle finger. This procedure will be performed on the right and left hand separately. The patient is instructed to judge if he/she felt a delay between the two vibratory bursts. The inner stimulus interval (ISI) is RECORDED when the participant indicates that they can feel a difference in time between the two vibrations. The ISI can range from 10ms-110 ms
Movement disorders unified Parkinson's rating scale (MDS-UPDRS) part 1 change from baseline to 24 months. | 24 months
  The MDS-UPDRS part 1 focuses on non-motor symptoms, such as dementia, depression, and psychosis. The total summed score ranges from 0-52 with higher scores indicating increased non-motor impairment.
Movement disorders unified Parkinson's rating scale (MDS-UPDRS) part 2 change from baseline to 24 months. | 24 months
  The MDS-UPDRS part 2 focuses on the patient's ability to perform daily motor activities including dressing, grooming, and using utensils. The total summed score ranges from 0-52 with higher scores indicating increased daily motor impairment.
Movement disorders unified Parkinson's rating scale (MDS-UPDRS) part 4 change from baseline to 24 months. | 24 months
  The MDS-UPDRS 4 focuses on Measures the complications of treatment, e.g. dyskinesias and motor fluctuations. The total summed score ranges from 0-24 with higher scores indicating increased motor complications.
Parkinson's disease cognitive functional rating scale (PD-CFRS) change from baseline to 24 months. | 24 months
  The PD-CFRS capture subjective daily functional cognitive decline among patients with Parkinson's disease over the past 2 weeks. The scale ranges from 0 to 24, with higher scores indicative of cognitive decline.
Parkinson's Disease-Cognitive Rating Scale (PDCRS) change from baseline to 24 months. | 24 months
  The PDCRS is a cognitive test designed to designed to cover the full spectrum of cognitive defects associated with Parkinson's Disease. The total test score ranges from 0 - 134, with higher scores indicating less cognitive impairment.
Parkinsons disease quality of life questionnaire-39 (PDQ-39) change from baseline to 24 months | 24 months
  The PD Quality of Life Questionnaire-39 (PDQ-39) is a self-report questionnaire that examines health related difficulties specific to PD in eight quality of life categories within the last month. Items are grouped into eight scales that are scored by expressing summed item scores as a percentage score ranging between 0 and 100, with higher % indicating more health problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States